CLINICAL TRIAL: NCT07086781
Title: Expediting Access to Autism Specific Intervention for Young Autistic Children Living in Rural North Carolina: a Pilot Study
Brief Title: Resources for Optimizing Outcomes in Toddlers on the Spectrum
Acronym: ROOTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Foundation of Hope for Research and Treatment of Mental Illness (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-1164
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Navigation (Experimental): Participants randomized to the Family Navigation condition will receive up to 4 research-based individual sessions with a trained navigator to support them in identifying and enrolling in recommended autism early intervention services. All navigation sessions will be delivered virtually via phone/Zoom.
  Interventions: Behavioral: Virtual Family Navigation
- Educational Materials (Active Comparator): The comparison condition ("Educational Materials") consists of providing the child's caregivers with information about early intervention and community-based supports (i.e., infant-toddler programs, transition to school-based supports, family support groups, local organizations). Families in this condition will receive this information throughout 4 timepoints in the first 3 months after enrolling.
  Interventions: Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Virtual Family Navigation — Participants randomized to the Family Navigation condition will receive up to 4 research-based individual sessions with a trained navigator to support them in identifying and enrolling in recommended autism early intervention services. All navigation sessions will be delivered virtually via phone/Zoom.
  Arms: Family Navigation
Behavioral: Educational Materials — The comparison condition ("Educational Materials") consists of providing the participant's caregivers information about early intervention and community-based supports (i.e., infant-toddler programs, transition to school-based supports, family support groups, local organizations. Families in this condition will receive this information throughout 4 timepoints in the first 3 months after enrolling.
  Arms: Educational Materials

SUMMARY:
The goal of this clinical trial is to assess whether telehealth-based Family Navigation (FN) expedites enrollment (e.g., reduces time in days) in community-based autism intervention for toddlers under the age of 4 living in Rural NC after their initial diagnosis of autism.

The main questions it aims to answer are:

Does Family Navigation decrease the time to initiation of intervention for rural toddlers with autism?

Does Family Navigation improve developmental outcomes at 18 months post-diagnosis of autism?

Does Family Navigation improve caregiver well-being?

Caregivers in the Family Navigation condition will receive 4 research-based individual sessions with a trained navigator to support them in identifying and enrolling in recommended autism early intervention services. All navigation sessions will be delivered virtually via phone/Zoom.

Researchers will compare participants who receive family navigation to participants who receive the standard of care (educational materials) to see if family navigation outperforms the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Children up to 48 months who have a new diagnosis of autism (within the last month) or who are waiting for a diagnosis of autism AND their caregiver.
* Live in North Carolina, in one of the 78 rural counties.
* Caregiver must be over the age of 18
* The caregiver must speak conversationally fluent English.

Exclusion Criteria:

* No access to a telephone or internet connection for phone calls or video conferencing.
* Diagnosis of autism spectrum disorder is ruled out in the child.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Time to initiation of autism specific intervention | Diagnosis to 18 months post
  The date of initiation (date 1) of autism-specific intervention will be the date that families report the first session with a therapist following the diagnosis (date 2). Time will be calculated as the number of days elapsed between these two dates (date 2 - date 1).

SECONDARY OUTCOMES:
Caregiver Well-Being Score | 6 months post diagnosis
  Scores on the General Well-Being Schedule will be used to measure caregiver well-being. Total scores range from 0-110. Higher scores are indicative of more positive well-being. There are 3 proposed scoring cut-points: 0-60 reflects "severe distress", 61-72 reflects "moderate distress", and 73-110 reflects "positive well-being). The investigators will compare means and standard deviations between groups.
Change in Raw Scores on Visual Reception domain of the MSEL | Baseline and 18 months post diagnosis
  This outcome will assess individual-level change in raw scores on the Mullen Scales of Early Learning (MSEL), Visual Reception domain. Raw scores will ne used instead of standard scores to detect meaningful change within-subject change. Standard scores in this population are known to exhibit floor effects in this population, which can obscure meaningful gains.
  Raw scores will be analyzed as continuous variables. The investigators will report change scores (follow-up minus baseline), individual trajectories, and summary statistics (mean, SD). Where appropriate, linear mixed-effects models or other growth modeling approaches will be used to account for within-subject variability.
  Higher scores on the MSEL indicate greater developmental progress. Raw scores on the Visual Reception domain range from 0-50.
Change in Raw Scores on Expressive Language domain of the MSEL | Baseline and 18 months post diagnosis
  This outcome will assess individual-level change in raw scores on the Mullen Scales of Early Learning (MSEL), Expressive Language domain. Raw scores will be used instead of standard scores to detect meaningful change within-subject change. Standard scores in this population are known to exhibit floor effects in this population, which can obscure meaningful gains.
  Raw scores will be analyzed as continuous variables. The investigators will report change scores (follow-up minus baseline), individual trajectories, and summary statistics (mean, SD). Where appropriate, linear mixed-effects models or other growth modeling approaches will be used to account for within-subject variability.
  Higher scores on the MSEL indicate greater developmental progress. Raw scores on the Expressive Language domain range from 0 - 50.
Change in Raw Scores on Receptive Language domain of the MSEL | Baseline and 18 months post diagnosis
  This outcome will assess individual-level change in raw scores on the Mullen Scales of Early Learning (MSEL), Receptive Language domain. Raw scores will be used instead of standard scores to detect meaningful change within-subject change. Standard scores in this population are known to exhibit floor effects in this population, which can obscure meaningful gains.
  Raw scores will be analyzed as continuous variables. The investigators will report change scores (follow-up minus baseline), individual trajectories, and summary statistics (mean, SD). Where appropriate, linear mixed-effects models or other growth modeling approaches will be used to account for within-subject variability.
  Higher scores on the MSEL indicate greater developmental progress. Raw scores on the Receptive Language domain range from 0 - 48.
Change in Raw Scores on Fine Motor domain of the MSEL | Baseline and 18 months post diagnosis
  This outcome will assess individual-level change in raw scores on the Mullen Scales of Early Learning (MSEL), Fine Motor domain. Raw scores will be used instead of standard scores to detect meaningful change within-subject change. Standard scores in this population are known to exhibit floor effects in this population, which can obscure meaningful gains.
  Raw scores will be analyzed as continuous variables. The investigators will report change scores (follow-up minus baseline), individual trajectories, and summary statistics (mean, SD). Where appropriate, linear mixed-effects models or other growth modeling approaches will be used to account for within-subject variability.
  Higher scores on the MSEL indicate greater developmental progress. Raw scores on the Visual Reception domain range from 0 - 49.
Change in Raw Scores on ABAS-3 Conceptual, Social and Practical Domains | Baseline and 18 months post diagnosis
  This outcome will assess change in raw scores for each of the three adaptive domains (Conceptual, Social and Practical) from the Adaptive Behavior Assessment System, Third Edition (ABAS-3). Raw scores offer greater sensitivity for detecting within-subject developmental changes over time. Each domain will be analyzed separately as a continuous variable. Where applicable, domain raw scores will also be summed to provide an exploratory composite.
  Higher scores indicate greater adaptive skill development.
  Conceptual domain raw score range: 0-222 Social domain raw score range: 0 - 144 Practical domain raw score range: 0-279

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Caravella, PhD, Principal Investigator — Carolina Institute for Developmental Disabilities
Locations (1):
- Carolina Institute for Developmental Disabilities, Carrboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator must have approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.